CLINICAL TRIAL: NCT03730142
Title: A Phase Ⅰ Study of PI3K/mTOR Dual Inhibitor WXFL10030390 to Evaluate the Safety, Tolerability and Pharmacokinetics in Patients With Advanced Solid Tumors or Lymphoma
Brief Title: A Study of WXFL10030390 in Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiatan Pharmatech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JYA0101
Record Dates: First submitted 2018-10-21; First posted 2018-11-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Advanced Cancer
Keywords: phosphoinositide-3 kinase (PI3K); mammalian target of rapamycin (mTOR)
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WXFL10030390 tablet (Experimental): WXFL10030390 continuous oral dosing (0.1 mg once a day)
  WXFL10030390 continuous oral dosing (0.2 mg once a day)
  WXFL10030390 continuous oral dosing (0.4 mg once a day)
  WXFL10030390 continuous oral dosing (0.7 mg once a day)
  WXFL10030390 continuous oral dosing (1.1 mg once a day)
  WXFL10030390 continuous oral dosing (1.4 mg once a day)
  WXFL10030390 continuous oral dosing (1.7 mg once a day)
  Interventions: Drug: WXFL10030390

INTERVENTIONS:
Drug: WXFL10030390 — WXFL10030390 is a tablet in the form of 0.1mg and 0.5mg, oral, once a day.
  Other Names: WX390

SUMMARY:
WXFL10030390 (WX390) is a novel oral small molecular that inhibits phosphoinositide-3 kinase (PI3K) and mammalian target of rapamycin (mTOR) and has demonstrated potent inhibitory effects on multiple human tumor xenografts. The first-in-human study is conducted to assess the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT), to evaluate the pharmacokinetics, safety and preliminary anti-tumor activity of WX390 at single dose and multiple doses.

DETAILED DESCRIPTION:
This study will be an open-lable, phase Ⅰ study and will evaluate the safety and pharmacokinetics of WX390 after a single administration followed by a 28-day continuous course of therapy; evaluate the safety and preliminary efficacy in an open-lable administration of WX390 at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 and ≤75 years of age
* Histological or cytological confirmed advanced solid tumor or lymphoma, standard regimen failed or no standard regimen available
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy of more than 3 months
* At least one measurable lesion according to RECIST 1.1 or Lugano 2014
* Adequate organic function: Absolute neutrophil count (ANC) ≥2.0×109/L，PLT≥100×109/L，Hb≥9g/L hepatic function:TBIL≤1.5×upper limit of normal (ULN)，Alanine aminotransferase (ALT) ≤2.5×ULN，aspartate aminotransferase (AST) ≤2.5×ULN; renal function:Cr≤1.5×ULN and>50ml/min; coagulation function: APTT≤1.5 ×ULN，PT≤1.5 ×ULN, INR≤1.5 ×ULN; GLU<7mmol/L and HbA1C<7%; TG≤1.5×ULN，CHOL≤1.5×ULN
* Subjects who have the fertility should agree to use reliable contraceptive methods during this study and subsequently at least 12 weeks after the last administration; for female subjects, the blood pregnancy test should be negative within 7 days prior to the enrollment
* Signed and dated informed consent

Exclusion Criteria:

* Anti-cancer therapy within 4 weeks prior to the initiation of investigational treatment
* Surgery within 4 weeks prior to the initiation of study treatment
* Use of strong inducers or inhibitors of CYP3A4 within 1 weeks before the first dose of study treatment. See Appendix 5 for a list of such medications
* Received corticosteroids treatment or other immunodepressant within 2 weeks before the first dose of study treatment
* Toxicity from a previous anti-tumor treatment that does not return to Grade 0 or 1 (except for alopecia)
* Patients with clinical symptomatic brain metastases, spinal compression, meningitis carcinomatosa or other evidence that shows uncontrolled brain or spinal metastases
* Previous treatment with PI3K/mTOR inhibitors
* Patients who once or being suffer Interstitial lung disease
* Evidence of ongoing or active infection
* History of human immunodeficiency virus (HIV) infection
* History of hepatitis B or C infection
* Clinically significant cardiovascular disease, including but not limited to acute coronary syndrome, congestive heart-failure, cerebral stroke within 6 months prior to enrollment, New York Heart Association Class ≥II cardiac functional grading or left ventricular ejection fraction (LVEF) < 50%
* Inability to take medication orally
* Severe gastrointestinal disease leading to diarrhea
* Diabetics receiving insulin treatment
* Patients with active autoimmune disease (including systemic lupus erythematosus, rheumatoid arthritis, nodular vasculitis)
* Abuse of alcohol or drugs
* People with cognitive and psychological abnormality or with low compliance
* Pregnant or lactating women
* Researchers believe that subjects may not be able to complete the study or may not be able to comply with the requirements of this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
Adverse Events evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | From first dose to within 30 days after the last dose
  The safety and tolerability of WXFL10030390 will be evaluated based on adverse events data. Other safety parameters include physical examination, clinical laboratory tests including coagulation function, renal function, hepatic function, blood glucose and blood lipid.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 28 days
  Cmax will be determined for an oral administration of WXFL10030390 tablets.
Time to reach plasma Cmax (tmax) | 28 days
  tmax will be determined for an oral administration of WXFL10030390 tablets.
Area under the plasma concentration-time curve (AUC) | 28 days
  AUC will be determined for an oral administration of WXFL10030390 tablets.
Terminal elimination half-life (t½) | 28 days
  t½ will be determined for an oral administration of WXFL10030390 tablets.
Recommended study Phase II dose (RP2D) | Up to 1 year
  The recommended phase 2 dose (RP2D) of WXFL10030390 will be determined based on pharmacokinetics, safety and tolerability, as well as preliminary efficacy.
Disease control rate | From first dose to within 30 days after the last dose
  The sum of complete responses (CR) + partial responses (PR) + stable disease (SD) as determined by Response Evaluation Criteria in Solid Tumors (RECIST) or Lugano 2014 criteria
Objective response rate | From first dose to within 30 days after the last dose
  Defined as complete response [CR] + partial response [PR]) as determined by Response Evaluation Criteria in Solid Tumors (RECIST) or Lugano 2014 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Doctor, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No